CLINICAL TRIAL: NCT03814109
Title: Randomized, Double-blind, Triple-dummy, National, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Leningrado Association in the Treatment of Hypertension
Brief Title: Efficacy and Safety of Leningrado Association in the Treatment of Hypertension
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0418 - LENINGRADO
Record Dates: First submitted 2019-01-22; First posted 2019-01-23 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Arterial Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — levamlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LENINGRADO (Experimental): The study is triple-dummy. Thus, the patient will take 3 tablets, as follow:
  1 tablet Leningrado association,1 tablet indapamide placebo, 1 tablet levamlodipine placebo, oral, once a day.
  Interventions: Drug: LENINGRADO association; Other: Indapamide SR Placebo; Other: Levamlodipine placebo
- Indapamide (Active Comparator): The study is triple-dummy. Thus, the patient will take 3 tablets, as follow:
  1 tablet indapamide 1,5 mg, 1 tablet Leningrado association placebo, and 1 tablet levamlodipine placebo, oral, once a day.
  Interventions: Drug: Indapamide SR 1.5 MG; Other: Leningrado association Placebo; Other: Levamlodipine placebo
- Levamlodipine (Active Comparator): The study is triple-dummy. Thus, the patient will take 3 tablets, as follow:
  1 tablet levamlodipine 2.5/ 5 mg, 1 tablet indapamide placebo, and 1 tablet Leningrado association placebo, oral, once a day.
  Interventions: Drug: Levamlodipine 2.5/ 5 mg; Other: Leningrado association Placebo; Other: Indapamide SR Placebo

INTERVENTIONS:
Drug: LENINGRADO association — 1 coated sustained-release tablet, oral, once a day.
  Other Names: EMS association
  Arms: LENINGRADO
Drug: Indapamide SR 1.5 MG — 1 coated sustained-release tablet, oral, once a day.
  Arms: Indapamide
Drug: Levamlodipine 2.5/ 5 mg — 1 tablet, oral, once a day.
  Arms: Levamlodipine
Other: Leningrado association Placebo — 1 coated sustained-release tablet, oral, once a day.
  Other Names: Placebo
  Arms: Indapamide; Levamlodipine
Other: Indapamide SR Placebo — 1 coated sustained-release tablet, oral, once a day.
  Other Names: Placebo
  Arms: LENINGRADO; Levamlodipine
Other: Levamlodipine placebo — 1 tablet, oral, once a day.
  Other Names: Placebo
  Arms: Indapamide; LENINGRADO

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Leningrado association on the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or more;
* Participants diagnosed with hypertension (mild to moderate), mild to moderate cardiovascular risk, not controlled by monotherapy and/ or lifestyle modification;

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* BP ≥ 180/110 mmHg;
* Participants with BMI (body mass index) ≥ 40 Kg/m2;
* Previous diagnosis of secondary hypertension;
* History of taget organ damage;
* History of cardiovascular, hepatic and renal disease;
* History of gout, diabetes mellitus and hypokalemia;
* Current medical history of cancer;
* Current smoking;
* History of alcohol abuse or drug use;
* Pregnancy or risk of pregnancy and lactating patients;
* Known allergy or hypersensitivity to the medicines components used during the clinical trial;
* Participation in clinical trial in the year prior to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure levels, as measured by 24h-ABPM at the initial visit and final visit. | 56 days

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study | 70 days